CLINICAL TRIAL: NCT03554070
Title: Thulium Fiber Laser Enucleation of the Prostate (ThuFLEP): Short-Term Efficacy and Safety Trial
Brief Title: Thulium Fiber Laser Enucleation of the Prostate (ThuFLEP): Efficacy and Safety
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: I.M. Sechenov First Moscow State Medical University (Other)
Responsible Party: Principal Investigator, Dmitry Enikeev, MD, PhD, Deputy Director for Science, I.M. Sechenov First Moscow State Medical University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Sechenov-ThuFLEP18
Record Dates: First submitted 2018-05-17; First posted 2018-06-12 (Actual); Last update posted 2021-07-22 (Actual); Status verified 2021-07

CONDITIONS: Prostatic Hyperplasia
Keywords: Prostate; BPH; Laser; Endoscopic Enucleation of the Prostate; Thulium; Thulium Fiber Laser
MeSH Terms: conditions — Prostatic Hyperplasia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Infravesical Obstruction (Experimental): Patients with infravesical obstruction due to BPH (IPSS > 20, Qmax < 10), who underwent Thulium Fiber Laser Enucleation of the Prostate.
  Interventions: Procedure: Thulium Fiber Laser Enucleation of the Prostate; Device: Thulium Fiber Laser "Urolase"

INTERVENTIONS:
Procedure: Thulium Fiber Laser Enucleation of the Prostate — Thulium laser enucleation of the prostate is performed using the two-lobe or en-bloc techniques. Incision depth is limited to the circular fibers of the prostate capsule. The left lobe is enucleated first, starting at the 5 o'clock position. The endoscope is then introduced counterclockwise at the 2 o'clock position. Next, an incision is made at 12 o'clock and extended to the level of the verumontanum. The incisions at the 12 and 2 o'clock positions are connected, and the left lobe is enucleated into the bladder. The right lobe of the gland is enucleated in a similar manner: the initial incision at 7 o'clock was made clockwise, an 11 o'clock incision is then extended along the capsule to join with the previous cut. The final step is morcellation of hyperplastic nodes.
Device: Thulium Fiber Laser "Urolase" — Urolase system (NTO IRE-POLUS, Russian Federation) is a thulium doped fiber laser.
  Max. power of 120 W and energy of 8 J. Wavelength - 1,94 µm, incision depth - 0,2 mm.

SUMMARY:
The aim of our study is to estimate the efficacy, safety and postoperative complications of the thulium fiber laser enucleation of the prostate (ThuFLEP) with Urolase system (NTO IRE-POLUS, Russia).

DETAILED DESCRIPTION:
In all patients, IPSS, Qmax, QoL, prostate volume, and IIEF-5 are measured prior to surgery.

For ThuFLEP, we use the Urolase system (NTO IRE-POLUS, Russia) and a 600 mcm fiber. The thulium fiber laser is set with a mean output power of 60 W and energy of 1.5 J. Tissue morcellation is completed with the Piranha Morcellator (Richard Wolf, Germany).

At the end of the procedure a 22 French three-way Foley catheter is placed. IPSS, Qmax, QoL, prostate volume are recorded at 1, 3 and 6 months after surgery. IIEF-5 are recorded at 3 and 6 months after surgery.

ELIGIBILITY:
Inclusion Criteria:

* Men aged 18 or older
* Infravesical obstruction due to prostatic hyperplasia (IPSS > 20 or Qmax <10)

Exclusion Criteria:

* Participation in another clinical study
* Prostate cancer (pathology confirmed)
* Urinary tract infection
* Neurogenic bladder

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 500 (Estimated)
Dates: Start 2018-03-01 (Actual); Primary Completion 2021-07-01 (Actual); Study Completion 2021-09-01 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline IPSS at 1,3 and 6 months | baseline and at 1,3 and 6 months
  International Prostate Symptom Score
Change from Baseline Qmax at 1,3 and 6 months | baseline and at 1,3 and 6 months
  Maximal urinary flow rate

SECONDARY OUTCOMES:
Change from Baseline QoL at 1,3 and 6 months | baseline and at 1,3 and 6 months
  Quality of Life (IPSS-QoL scale)
Change from Baseline IIEF-5 at 3 and 6 months | baseline and at 3 and 6 months
  The International Index of Erectile Function - 5
Change from Baseline Prostate Volume at 1,3 and 6 months | baseline and at 1,3 and 6 months
  Prostate volume measured by ultrasound (transrectal or abdominal)

CONTACTS AND LOCATIONS:
Overall Officials: Dmitry Enikeev, Study Director — I.M. Sechenov First Moscow State Medical University
Locations (1):
- Clinic of Urology, I.M. Sechenov First Moscow State Medical University, Moscow, Russia

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Enikeev D, Glybochko P, Okhunov Z, Alyaev Y, Rapoport L, Tsarichenko D, Enikeev M, Sorokin N, Dymov A, Taratkin M. Retrospective Analysis of Short-Term Outcomes After Monopolar Versus Laser Endoscopic Enucleation of the Prostate: A Single Center Experience. J Endourol. 2018 May;32(5):417-423. doi: 10.1089/end.2017.0898. Epub 2018 Mar 13. PMID 29430969
- [Background] Glybochko PV, Rapoport LM, Enikeev ME, Enikeev DV. Holmium laser enucleation of the prostate (HoLEP) for small, large and giant prostatic hyperplasia: tips and tricks. Urologia. 2017 Aug 1;84(3):169-173. doi: 10.5301/uj.5000232. Epub 2017 May 10. PMID 28497447